CLINICAL TRIAL: NCT02561559
Title: Phase II Study to Evaluate Feasibility and Safety of Stereotactic Body Radiation Radiotherapy (SBRT) for Lung Metastases From Soft Tissue Sarcoma
Brief Title: SBRT Treatment for Lung Metastasis From Soft Tissue Sarcoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Other Study IDs: 1393
Record Dates: First submitted 2015-09-25; First posted 2015-09-28 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Metastasis From Malignant Tumor of Soft Tissues

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lung metastasis from soft-tissue sarcoma: Lung metastases from soft-tissue sarcoma
  Interventions: Radiation: Lung metastasis from soft-tissue sarcoma

INTERVENTIONS:
Radiation: Lung metastasis from soft-tissue sarcoma — Tretament based on Intensity Modulated Radiation Therapy (IMRT) using Volumetric Modulated Arc Therapy (VMAT)

SUMMARY:
In this study the investigators treat PM oligometastatic patients with SBRT. Our objective is to evaluate rate of local control of treated lesions in patients treated with Intensity Modulated Radiation Therapy (IMRT) using Volumetric Modulated Arc Therapy (VMAT) for lung metastases from STS.

DETAILED DESCRIPTION:
The investigators started to treat PM oligometastatic patients with Stereotactic Body Radiotherapy.

The investigators objective is to evaluate rate of local control of treated lesions in patients treated with Intensity Modulated Radiation Therapy (IMRT) using Volumetric Modulated Arc Therapy (VMAT) for lung metastases from soft-tissue sarcomas. Overall and disease free survival will be evaluated as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 anni -85 years
* PS according to ECOG 0-2
* Histopathologically confirmation of soft tissue sarcoma
* Metastatic lung lesion less than 4
* Controlled primary tumor and other metastatic lesions
* Metastatic lesion less than 5 such as the definition of oligometastatic patients
* Written informed consent
* Contraindication to surgical resection
* Estimated survival ≥ 3 months
* Absence of progressive disease longer than 6 months
* No chemotherapy was given for at least 3 months after SBRT
* Maximum diameter ≤ 5 cm

Exclusion Criteria:

* Prior thorax radiation therapy
* Age > 85 years
* PS according to ECOG >2
* Pregnant women
* Maximum diameter ≥ 5.1 cm
* Total volume of lung lesion greater than 1/3 of the whole pulmonary parenchima

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients affected by soft-tissue sarcomas with lung metastases unsuitable for surgery
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Local control of treated lesions | 12 months
  Evaluation of proportion of patients free from progression from starting radiotherapy

SECONDARY OUTCOMES:
Overall survival of treated patients | 4 years
  Evaluation of proportion of patients alive
Disease free survival of treated patients | 4 years
  Evaluation of proportion of patients alive and free from progression

CONTACTS AND LOCATIONS:
Overall Officials: Marta Scorsetti, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Milan, Italy

REFERENCES:
- [Background] Navarria P, Ascolese AM, Cozzi L, Tomatis S, D'Agostino GR, De Rose F, De Sanctis R, Marrari A, Santoro A, Fogliata A, Cariboni U, Alloisio M, Quagliuolo V, Scorsetti M. Stereotactic body radiation therapy for lung metastases from soft tissue sarcoma. Eur J Cancer. 2015 Mar;51(5):668-74. doi: 10.1016/j.ejca.2015.01.061. Epub 2015 Feb 13. PMID 25686482